CLINICAL TRIAL: NCT02120677
Title: A Pilot Study Investigating Antitumorigenic Potential of Topical Itraconazole in the Treatment of Basal Cell Carcinoma
Brief Title: Topical Itraconazole in the Treatment of Basal Cell Carcinoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00077461
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Basal Cell Carcinoma
Keywords: skin cancer; basal cell carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Itraconazole ointment (Experimental): Patients with histologically proven BCC will be eligible for study enrollment. 50% itraconazole compounded in petrolatum jelly will be applied under occlusion for up to 3 to 7 days.
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — Itraconazole comes in the form of capsules and liquid (oral solution). It is FDA approved for treatment of systemic Blastomycosis, Histoplasmosis and Aspergillosis in immunocompromised and non-immunocompromised patients at doses ranging from 200mg to 400mg daily. The current FDA approved dosage recommendation for treating toenail onychomycosis (nail fungus) is 200mg PO per day for 3 months. Test materials in this study will be prepared as an ointment (compounded in petrolatum jelly).
  Other Names: Sporanox

SUMMARY:
This research is being done to study the molecular effects of topically applied itraconazole ointment on the growth of basal cell carcinomas.

DETAILED DESCRIPTION:
Basal cell carcinoma is the most common type of skin cancer in Caucasians worldwide. Although rarely metastatic, it can be locally destructive causing disfigurement and pain. Current therapies include surgical removal, local destruction, radiotherapy and others.

Advances in understanding the molecular basis behind BCCs indicate that mutations in the hedgehog signaling pathway can lead to the development of many sporadically occurring basal cell carcinomas (BCCs). An oral drug that targets the hedgehog signaling pathway has been shown to be effective in treating patients with metastatic and inoperable BCCs. There is evidence that itraconazole, a commonly prescribed antifungal medication may also affect this pathway. It is not known whether itraconazole ointment applied topically can affect the growth of BCCs.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be over the age of 18 years
* Male
* Women who do not have child-bearing potential (history of hysterectomy, post-menopausal)
* Have a biopsy confirmed BCC that measures at least 6mm in size at the time of the initial evaluation (visit #1);
* Participant must be willing and comply with the requirements of the protocol;
* Participant must have the ability to understand and communicate with the investigator;
* Participant must provide informed consent.

Exclusion Criteria:

* Subject with significant congestive heart failure (CHF) or history of CHF, chronic renal failure, hepatic failure, neuropathy
* Subject with current skin diseases that the investigator feels is not safe for study participation including but not limited to severe atopic dermatitis, cutaneous T-cell lymphoma, erythroderma;
* Subjects on systemic medications known to affect the Hedgehog pathway (see Appendix I)
* Subjects on cisapride, oral midazolam, nisoldipine, felodipine, pimozide, quinidine, dofetilide, triazolam, methadone, levacetylmethadol (levomethadyl), lovastatin, simvastatin, dihydroergotamine, ergometrine (ergonovine), ergotamine and methylergometrine (methylergonovine), cisapride, pimozide, methadone, levacetylmethadol (levomethadyl), quinidine
* Subjects with history of hypersensitivity to azoles
* Subjects with Gorlin syndrome
* Subjects on chronic immunosuppression, or who have a history of compromised immune function (e.g. history of or current malignancy other than BCC/squamous cell skin cancers)
* Subjects who do not speak English or have difficulty hearing or are otherwise impaired for providing informed consent and communicating with the investigator;
* Subjects with a history of keloids or excessive scarring;
* Subjects with known allergy to lidocaine, epinephrine, itraconazole or petrolatum
* Women of child-bearing age/potential and/or able to conceive

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Downregulation in glucagon-like immunoreactivity (GLI) expression | Day 8
  We will report the proportion of patients by treatment cohort and overall that had a significant downregulation in GLI.

SECONDARY OUTCOMES:
Incidence, timing, and severity of treatment adverse events | 45 days
  Data on adverse events will be collected and reported by treatment cohort and overall.

CONTACTS AND LOCATIONS:
Overall Officials: Nikki Tang, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Department of Dermatology, Baltimore, Maryland, United States